CLINICAL TRIAL: NCT00779844
Title: Intravenous Anesthesia in Obese Patients: Propofol and Remifentanil Requirements
Brief Title: Anesthesic Propofol and Remifentanil Requirements in Obese Patients
Acronym: LoopObese
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: difficulty in recruiting
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008/02
Record Dates: First submitted 2008-10-23; First posted 2008-10-24 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Anesthesia; Obesity
Keywords: Anesthesia; Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): obese patients
  Interventions: Procedure: bariatric coelioscopic surgical procedure
- 2 (Active Comparator): lean patients
  Interventions: Procedure: supra-umbilical coelioscopic surgical procedure

INTERVENTIONS:
Procedure: bariatric coelioscopic surgical procedure — total intra-venous anesthesia (propofol and remifentanil) being delivered using a close-loop system with the Bispectral Index as the single input for the controller
  Arms: 1
Procedure: supra-umbilical coelioscopic surgical procedure — total intra-venous anesthesia (propofol and remifentanil) being delivered using a closed-loop system with the Bispectral Index as the single input for the controller
  Arms: 2

SUMMARY:
Pharmacokinetic models for anesthetic agents are questionable. The objective of the study is to compare the propofol and remifentanil doses required to maintain the bispectral index in the range 40-60 in two groups of patients: obese patients and lean patients

ELIGIBILITY:
Inclusion Criteria:

- Patients scheduled for a bariatric coelioscopic surgical procedure (obese patients) or for an upper abdominal laparoscopic procedure (lean patients)

Exclusion Criteria:

* age lower than 18 years,
* pregnant woman,
* presence of a central neurological disorder or a lesion cerebral, of a severe respiratory or hepatic insufficiency,
* allergy to propofol, or to soja or to peanuts, or to sufentanil, or to remifentanil, or to morphine, or to a muscle myorelaxant, or to an excipient,
* hypersensibility to sufentanil, or to remifentanil or to another derivate of fentanyl,
* allergy to latex,
* presence of a symptomatic gastroesophageal reflux,
* patients receiving a psychotropic treatment or a agonist-antagonist opiate,
* presence of predictive signs of difficult mask ventilation of difficult intubation (else than obesity)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2008-12; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Dose of propofol administered | intraoperatively

SECONDARY OUTCOMES:
remifentanil requirement, hemodynamic profile, time to extubation, performances of the automated system of propofol and remifentanil deliver | intraoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Marc Fischler, MD, Study Chair — Hopital Foch
Locations (1):
- Hôpital Européen Georges Pompidou, Paris, France

REFERENCES:
- [Background] Liu N, Chazot T, Genty A, Landais A, Restoux A, McGee K, Laloe PA, Trillat B, Barvais L, Fischler M. Titration of propofol for anesthetic induction and maintenance guided by the bispectral index: closed-loop versus manual control: a prospective, randomized, multicenter study. Anesthesiology. 2006 Apr;104(4):686-95. doi: 10.1097/00000542-200604000-00012. PMID 16571963
- [Background] Servin F, Farinotti R, Haberer JP, Desmonts JM. Propofol infusion for maintenance of anesthesia in morbidly obese patients receiving nitrous oxide. A clinical and pharmacokinetic study. Anesthesiology. 1993 Apr;78(4):657-65. doi: 10.1097/00000542-199304000-00008. PMID 8466066
- [Derived] Liu N, Lory C, Assenzo V, Cocard V, Chazot T, Le Guen M, Sessler DI, Journois D, Fischler M. Feasibility of closed-loop co-administration of propofol and remifentanil guided by the bispectral index in obese patients: a prospective cohort comparison. Br J Anaesth. 2015 Apr;114(4):605-14. doi: 10.1093/bja/aeu401. Epub 2014 Dec 10. PMID 25500680